CLINICAL TRIAL: NCT02612831
Title: Bariatric Surgery for Obese Patients With Chronic Renal Insufficiency
Acronym: BOKID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14APN01; 2014-A011884-43 (Other: ANSM)
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Disease; Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early bariatric surgery (Other): patient receive their procedure early (within 3 months)
  Interventions: Procedure: Early bariatric surgery
- Delayed bariatric surgery (Other): Patient receive their procedure later (in 12 - 15 months), following a year of optimal medical treatment
  Interventions: Procedure: Delayed bariatric surgery

INTERVENTIONS:
Procedure: Early bariatric surgery
  Arms: Early bariatric surgery
Procedure: Delayed bariatric surgery
  Arms: Delayed bariatric surgery

SUMMARY:
The creatinine clearance will be measured using two consecutive 24 hour urine collections, with the objective of minimizing errors due to poor quality urine collection.

The GFR will be measured by a reference method, because its estimation from blood creatinine levels (eGFR) by the MDRD study formula may be confounded by variations in muscle mass, and therefore creatinine production, following bariatric surgery. The method will remain the same in each center, and therefore consistent for any given patient, throughout the duration of the study. The GFR measurements will be performed after stopping any medication blocking the RAAS, and reducing diuretics for one week, with the introduction or increase of alpha-blockers or centrally-acting hypotensive agents. If it is impossible to stop RAAS-blockade (heart failure), the dose will at least be reduced for one week. This precaution is required to minimize the bias of functional renal insufficiency because the state of extracellular hydration is difficult to assess in obese subjects. Subsequent measurements of GFR will be performed in the same way.

The choice of the tracer to measure GFR may vary according to study center. 51Cr-EDTA, 99Tc-DTPA, iohexol or inulin may all be utilized. Because the assessment of edema is hazardous in extremely obese patients and because kidney disease favors edema formation, the simplified single injection method and the determination of plasma clearance measurement of the tracer is not reliable . Only the constant infusion method will be used to measure GFR. Briefly, GFR will be determined by calculating the glomerular clearance (Cl) from plasma concentrations (P) and renal excretions per unit of time (UxV) during infusion at a constant plasma level of the tracer (Cl=UxV/P). The result will be given as mean value of several consecutive clearances. Because correct urine collection is key for the procedure, seven collection periods (instead of 5 usually) will be performed for the calculation of the mean clearance. Bladder catheterization will be used only when it can be anticipated that the patient will not void satisfactorily. In the last 30 consecutive patients with mGFR below 60 ml/min/1,73m2, this occurred twice and the subjects were 70 and 79 years old. Therefore, this might occur exceptionably in the study. Raw data from each center will be sent to the coordination center (Nice) to examine and validate the calculation of mean clearance values. To that aim, extreme and non-representative clearances will be excluded. At least 3 of the 7 periods will be taken into account to calculate the mean values. For instance, in the last 30 consecutive patients with mGFR below 60 ml/min/1,73m2, investigators considered on average 4.7 periods and obtained a mean non-indexed GFR value of 40,7 ± 2,5 ml/min.

Primary assessment will be performed at one year, as a previous study has already suggested a significant benefit within this period [66], and because surgery can't be delayed further in these patients strongly expecting the intervention, but follow-up will be extended to three years or until the end of the study, in order to document whether the initial benefits of surgical intervention are maintained.

* A reduction in the absolute value of measured GFR (mGFR) following bariatric surgery is expected in the first six months after surgery (M0 - M6). However, the weight loss may allow an increased in mGFR indexed to body surface area up until M6, and above all towards M12.
* the investigators expect a subsequent stabilization of mGFR between M12 and M36 in the bariatric surgery group, and will seek to measure the anticipated reduction in mGFR in the control group who remain in a state of glomerular hyperfiltration.

All relevant cardiovascular, metabolic and nutritional parameters necessary to study the risk/benefit ratio of the intervention will be analyzed.

* Primary: bariatric surgery slows the progression of chronic kidney disease in the obese.
* Secondary: bariatric surgery improves survival, cardiovascular prognosis, metabolic, nutritional and inflammatory parameters, quality of life, and access to transplantation in the sub-group of patients whose GFR < 20ml/min/1.73m2 at inclusion, and there could be a chance loss for the patients in delaying surgery by one year.

ELIGIBILITY:
Inclusion Criteria:

* • patients aged 18 to 75 years;

  * obese with BMI ≥ 35 kg/m2 , despite at least six months of appropriate medical, nutritional, dietetic and psychotherapeutic management;
  * having received accurate information about the surgery and requesting the procedure;
  * considered eligible for bariatric surgery following discussion at the multi-disciplinary meeting;
  * having understood and accepted the need for long-term medical and surgical follow-up;
  * with a GFR estimated by MDRD < 60 ml/min/1,73 m2 ;
  * women of child-bearing age must be using an effective method of contraception;
  * valid status in the social security system;
  * having signed the informed consent document, included the care contract.

Exclusion Criteria:

* • patients on dialysis or with renal grafts,

  * estimated GFR < 15 ml/min/1,73m2 if proteinuria > 3 g/g of creatinuria,
  * progressive pathology with a life expectancy less than one year,
  * mental incapacity or severe mental illness,
  * severe, uncontrolled eating disorder,
  * pregnancy or breastfeeding,
  * alcohol or drug dependence.
  * Adults of the age of majority subject to guardianship court order or deprived of liberty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
change in mGFR medical treatment for chronic kidney disease with or without bariatric surgery using gastric bypass surgery or longitudinal gastrectomy . | 12 months
  The change in mGFR is calculated as the difference between mGFR at M12 and mGFR at M0. These differences will be compared between the groups using covariance analysis adjusted on initial mGFR values (M0). Additional adjustment will include variables described in the analysis strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology department, CHU de NICE, Nice, France